CLINICAL TRIAL: NCT01516827
Title: Effectiveness of Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) for Children With Post-traumatic Stress Disorder
Brief Title: Effectiveness of Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) for Children With Post-traumatic Stress Disorder (TreatChildTrauma)
Acronym: TCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Lutz Goldbeck, Head of Section for Psychotherapy Re-search and Behavioural Medicine, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCT-001-ULM
Record Dates: First submitted 2011-12-13; First posted 2012-01-25 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Children and Adolescents; Post-Traumatic Stress Disorder in Children and Adolescents
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TF-CBT (Experimental): 12 Sessions Trauma-focused Cognitive Behavioral Therapy including the child/adolescents and a non-abusive caregiver according to the treatment manual:
  Cohen JA, Mannarino AP, and Deblinger E (2006) Treating Trauma and Traumatic Grief in Children and Adolenscents. Guilford, N.Y.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)
- Wait-list (No Intervention): Patients in the control condition will be assigned to a wait-list (duration 4 months). During waiting time, clinical services will be provided as needed (excluding TF-CBT).

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) — TF-CBT (see also HThttp://tfcbt.musc.eduTH) is a manualised intervention for traumatized children and adolescents 7 to 16 years old and their parent/caregiver. The primary components are summarized by the acronym PRACTICE: Parenting skills, Psychoeducation, Relaxation, Affect modulation, Cognitive processing, Trauma narrative, In vivo mastery of trauma reminders, Conjoint child-parent session, and Enhancing safety and future development. We will use the manual as provided by Cohen et al. and available in German. The treatment program will comprise 12 sessions with children and parents (partly separated, partly conjoined sessions) of 90 minutes each. The 12 sessions will be distributed over a duration of 16 weeks.
  Arms: TF-CBT

SUMMARY:
This multi-site randomized controlled trial compares the effectiveness of Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) as developed by Cohen, Mannarino & Deblinger (2006) with a wait-list condition in a population of children aged 7-16 years who were exposed to traumatic events beyond the age of three years, at least three months ago, and developed Posttraumatic Stress Disorder (PTSD). Primary aims are to provide evidence that TF-CBT exceeds spontaneous remission of posttraumatic stress symptoms and to assess maintenance of treatment gains at 6 and 12 months post-treatment. Secondary aims are to evaluate the effectiveness of TF-CBT in reducing other psychopathology and cognitive distortions of patients and caregivers and to explore moderators and mediators of treatment response. The trial will contribute to implement an evidence-based treatment for traumatized children across a variety of healthcare settings in Germany. The novel aspect is to evaluate the effectiveness of TF-CBT with a broad range of traumatized "real-world" patients in the context of the German mental healthcare system.

DETAILED DESCRIPTION:
Complete study protocol (in German) available from the PI lutz.goldbeck@uniklinik-ulm.de

ELIGIBILITY:
Inclusion Criteria:

* Age 7-16 years
* Exposure to a traumatic event (index trauma) after the age of 3 years, at least 3 months before assessment
* ≥35 points on the Clinician -Administered PTSD Scale for Children and Adolescents (CAPS-CA) total symptom severity score and at least one symptom per PTSD cluster related to the index trauma according to DSM IV diagnostic criteria
* PTSD should be the main mental health problem, patients with co-morbid mental disorders are included
* No major brain injury of the child due to the traumatic event (Glasgow Coma Scale <9 points at primary medical examination)
* Co-operation of at least one non-offending primary caregiver (improves treatment outcome)
* Living within reasonable distance (max 1 hour of travel) to the treatment center to allow treatment on a weekly basis (feasibility)

Exclusion Criteria:

* Psychosis
* Acute suicidality
* Psychopharmacological medication started or changed up to 6 weeks before first assessment

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-Administered PTSD Scale for Children and Adolescents (CAPS-CA) | Change from Baseline at 16 weeks (=end of treatment)
  Symptom severity score

SECONDARY OUTCOMES:
Change from Baseline in Schedule for Affective Disorders and Schizophrenia for School Aged Children (K-SADS-PL) | Change from Baseline at 16 weeks (=end of treatment)
  change in co-morbid psychiatric disorders
Change from Baseline in Children's Global Assessment Scale (CGAS) | Change from Baseline at 16 weeks (=end of treatment)
  Global impairment
Change from Baseline in UCLA PTSD Reaction Index (self-report and caregiver report) | Change from Baseline at 8 weeks (=mid-treatment)
  Post-traumatic stress symptoms
Change from Baseline in Self-report for childhood anxiety related disorders (SCARED; Self-report and caregiver report) | Change from Baseline at 8 weeks (=mid-treatment)
  Anxiety
Change from Baseline in Children's Depression Inventory (CDI) | Change from Baseline at 8 weeks (=mid-treatment)
  Depression
Change from Baseline in Child Behavior Checklist (CBCL 4/18) | Change from Baseline at 8 weeks (=mid-treatment)
  General Psychopathology
Change from Baseline in Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen (ILK; Self-report and caregiver report) | Change from Baseline at 8 weeks (=mid-treatment)
  Quality of Life
Change from Baseline in Child Post Traumatic Cognitions Inventory (CPTCI) | Change from Baseline at 8 weeks (=mid-treatment)
  Trauma-related Cognitions (Child)
Change from Baseline in The Posttraumatic Cognitions Inventory (PTCI) | Change from Baseline at 8 weeks (=mid-treatment)
  Trauma-related cognitions (Parent)
Change from Baseline in Posttraumatic Diagnostic Scale (PDS) | Change from Baseline at 8 weeks (=mid-treatment)
  Parental symptoms: PTSD
Change from Baseline in Beck Depression Inventory (BDI-II) | Change from Baseline at 8 weeks (=mid-treatment)
  Parental Symptoms: Depression
Change from Baseline in State-Trait-Anxiety-Inventory (STAI) | Change from Baseline at 8 weeks (=mid-treatment)
  Parental symptoms: Anxiety
Change from Baseline in Children's Global Assessment Scale (CGAS) | Change from Baseline at 6 months post-treatment
  Global impairment
Change from Baseline in Children's Global Assessment Scale (CGAS) | Change from Baseline at 12 months post-treatment
  Global impairment
Change from Baseline in UCLA PTSD Reaction Index (self-report and caregiver report) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in UCLA PTSD Reaction Index (self-report and caregiver report) | Change rom Baseline at 6 months post-treatment
Change from Baseline in UCLA PTSD Reaction Index (self-report and caregiver report) | Change from baseline at 12 months post-treatment
Change from Baseline in Self-report for childhood anxiety related disorders (SCARED; Self-report and caregiver report) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Self-report for childhood anxiety related disorders (SCARED; Self-report and caregiver report) | Change from Baseline at 6 months post-treatment
Change from Baseline in Self-report for childhood anxiety related disorders (SCARED; Self-report and caregiver report) | Change from Baseline at 12 months post-treatment
Change from Baseline in Children's Depression Inventory (CDI) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Children's Depression Inventory (CDI) | Change from Baseline at 6 months post-treatment
Change from Baseline in Children's Depression Inventory (CDI) | Change from Baseline at 12 months post-treatment
Change from Baseline in Child Behavior Checklist (CBCL 4/18) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Child Behavior Checklist (CBCL 4/18) | Change from Baseline at 6 months post-treatment
Change from Baseline in Child Behavior Checklist (CBCL 4/18) | Change from Baseline at 12 months post-treatment
Change from Baseline in Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen (ILK; Self-report and caregiver report) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen (ILK; Self-report and caregiver report) | Change from Baseline at 6 months post-treatment
Change from Baseline in Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen (ILK; Self-report and caregiver report) | Change from Baseline at 12 months post-treatment
Change from Baseline in Child Post Traumatic Cognitions Inventory (CPTCI) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Child Post Traumatic Cognitions Inventory (CPTCI) | Change from Baseline at 6 months post-treatment
Change from Baseline in Child Post Traumatic Cognitions Inventory (CPTCI) | Change from Baseline at 12 months post-treatment
Change from Baseline in The Posttraumatic Cognitions Inventory (PTCI) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in The Posttraumatic Cognitions Inventory (PTCI) | Change from Baseline at 6 months post-treatment
Change from Baseline in The Posttraumatic Cognitions Inventory (PTCI) | Change from Baseline at 12 months post-treatment
Change from Baseline in Posttraumatic Diagnostic Scale (PDS) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Posttraumatic Diagnostic Scale (PDS) | Change from Baseline at 6 months post-treatment
Change from Baseline in Posttraumatic Diagnostic Scale (PDS) | Change from Baseline at 12 months post-treatment
Change from Baseline in Beck Depression Inventory (BDI-II) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in Beck Depression Inventory (BDI-II) | Change from Baseline at 6 months post-treatment
Change from Baseline in Beck Depression Inventory (BDI-II) | Change from Baseline at 12 months post-treatment
Change from Baseline in State-Trait-Anxiety-Inventory (STAI) | Change from Baseline at 16 weeks (=end of treatment)
Change from Baseline in State-Trait-Anxiety-Inventory (STAI) | Change from Baseline at 6 months post-treatment
Change from Baseline in State-Trait-Anxiety-Inventory (STAI) | Change from Baseline at 12 months post-treatment
Change from baselinein Clinician-Administered PTSD Scale for Children and Adolescents (CAPS-CA) | Change from Baseline at 6 monts post-treatment
  Symptom severity score
Change from Baseline in Clinician-Administered PTSD Scale for Children and Adolescents (CAPS-CA) | Change from baseline at 12 months post-treatment
  Symptom severity score

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Goldbeck, Ph.D., Principal Investigator — University Ulm
Locations (8):
- Germany (8):
  - Vivantes Klinik für Kinder- und Jugendpsychiatrie, Psychotherapie und Psychosomatik, Berlin
  - Vestische Kinder- und Jugendklinik Datteln, Datteln
  - Psychiatrische Klinik Lüneburg, Lüneburg
  - Klinik für Psychiatrie und Psychotherapie, Mannheim
  - Traumaambulanz LMU, München
  - ZfP Südwürttemberg Weissenau, Ravensburg
  - Klinik für Kinder- und Jugendpsychiatrie und -psychotherapie, Saarbrücken
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Tutus D, Pfeiffer E, Plener PL, Rosner R, Bernheim D, Sachser C. The Change in Parental Symptoms and Dysfunctional Cognitions in the Course of Trauma-Focused Cognitive-Behavioral Therapy: Sustainability Until One-Year Post-Treatment. J Child Adolesc Psychopharmacol. 2021 Mar;31(2):129-136. doi: 10.1089/cap.2020.0097. Epub 2020 Dec 23. PMID 33370208
- [Derived] Lindebo Knutsen M, Sachser C, Holt T, Goldbeck L, Jensen TK. Trajectories and possible predictors of treatment outcome for youth receiving trauma-focused cognitive behavioral therapy. Psychol Trauma. 2020 May;12(4):336-346. doi: 10.1037/tra0000482. Epub 2019 Jul 25. PMID 31343205
- [Derived] Tutus D, Goldbeck L, Pfeiffer E, Sachser C, Plener PL. Parental dysfunctional posttraumatic cognitions in trauma-focused cognitive behavioral therapy for children and adolescents. Psychol Trauma. 2019 Oct;11(7):722-731. doi: 10.1037/tra0000419. Epub 2018 Dec 20. PMID 30570287
- [Derived] Sachser C, Keller F, Goldbeck L. Complex PTSD as proposed for ICD-11: validation of a new disorder in children and adolescents and their response to Trauma-Focused Cognitive Behavioral Therapy. J Child Psychol Psychiatry. 2017 Feb;58(2):160-168. doi: 10.1111/jcpp.12640. Epub 2016 Sep 28. PMID 27677771
- [Derived] Unterhitzenberger J, Eberle-Sejari R, Rassenhofer M, Sukale T, Rosner R, Goldbeck L. Trauma-focused cognitive behavioral therapy with unaccompanied refugee minors: a case series. BMC Psychiatry. 2015 Oct 23;15:260. doi: 10.1186/s12888-015-0645-0. PMID 26497391